CLINICAL TRIAL: NCT00667407
Title: A Randomized, Double-Blind Study to Determine the Efficacy of Levalbuterol Versus Racemic Albuterol in the Treatment of Acute Asthma
Brief Title: Efficacy and Safety of Levalbuterol Versus Racemic Albuterol in Asthma
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sumitomo Pharma America, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 051-915
Record Dates: First submitted 2008-04-24; First posted 2008-04-28 (Estimated); Last update posted 2012-02-22 (Estimated); Status verified 2012-02

CONDITIONS: Asthma
Keywords: Asthma
MeSH Terms: conditions — Asthma | interventions — Levalbuterol

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Levalbuterol 1.25 mg
  Interventions: Drug: Levalbuterol 1.25 mg
- 2 (Active Comparator): Racemic Albuterol 2.5 mg
  Interventions: Drug: Racemic Albuterol Sulfate

INTERVENTIONS:
Drug: Levalbuterol 1.25 mg — levalbuterol 1.25 mg Period I: administered every 20 minutes for the first 3 doses, and then every 40 minutes for the next 3 doses; then as clinically indicated.
  Period II: TID for 3 days (same time of day), then PRN to TID for 7 days
  Other Names: Xopenex HCl Inhalation Solution
  Arms: 1
Drug: Racemic Albuterol Sulfate — Racemic Albuterol 2.5 mg Period I: every 20 min for the first 3 doses, then every 40 min for the next 3 doses, then as clinically indicated.
  Period II: TID for 3 days then PRN to TID for 7 days
  Other Names: Ventolin Inhalation Solution
  Arms: 2

SUMMARY:
To investigate the Efficacy and Safety of Levalbuterol versus Racemic Albuterol in the Treatment of Acute Asthma.

DETAILED DESCRIPTION:
This study is a double-blind, randomized, active-controlled, multicenter, parallel-group trial of levalbuterol in adult subjects with acute reversible airways disease. Approximately 600 subjects will be enrolled and study participation will consist of 2 periods: Period I (Acute Period): Double-blind treatment in the Emergency Department (ED) or Clinic until disposition, for a maximum of 24 hours of double-blind treatment and Period II (Post-Acute Period): Subjects discharged from the ED or Clinic will continue double blind treatment (with the same treatment provided as rescue medication as MDI) for approximately 10 days. Subjects will be contacted by telephone 30 days post discharge to assess relapse. This study was previously posted by Sepracor Inc. In October 2009, Sepracor Inc. was acquired by Dainippon Sumitomo Pharma., and in October 2010, Sepracor Inc's name was changed to Sunovion Pharmaceuticals Inc.

ELIGIBILITY:
Inclusion Criteria:

* Male and female subjects must be at least greater than or equal to 18 years of age at the time of consent.
* Subjects must have history of asthma for at least 6 months.
* Subjects must present to the emergency department (ED) or clinic with forced expiratory volume in one second (FEV1) of 20 to 55% (inclusive) predicted at baseline
* Subjects must have O2 saturation greater than or equal to 90% at room air or with no more than 6 Liters/minute supplemental oxygen and no other cause of wheezing or shortness of breath other than asthma as determined by the physician.
* Prior use of a beta-agonist (e.g., Primatine Mist, albuterol, salmeterol, etc.) within 24 hours of presentation to the ED or Clinic.
* Smoked ≤ 10 pack-years or non-smoker.
* Be in good health with the exception of asthma and not suffering from any chronic condition which might affect their lung function, such as COPD or emphysema.
* Near-normal activity level between exacerbations.
* Subjects who are taking inhaled or systemic corticosteroids must be on a stable dose for at least 21 days prior to study entry.

Exclusion Criteria:

* Subjects who have received treatment for asthma in an ED, Clinic, or Urgent Care Center within 2 weeks prior to study entry.
* Based upon history or physical exam in the ED or Clinic, subjects with known or suspected cause of pulmonary symptoms other than asthma, such as COPD, CHF, pneumonia, pulmonary embolism, or angioedema.
* Subjects with a history of asthma episodes associated with hypercapnia, respiratory arrest, hypoxic seizures, or requiring intubation within 12 months prior to entry.
* Hospitalization for asthma within two months prior to entry.
* Female subjects who are pregnant or lactating.
* Subjects who have a history of a clinically significant psychiatric disorder within the last 3 months, with the exception of mild depression.
* Subjects who have participated in an investigational drug study within 30 days of study entry or have previously participated in the current trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 627 (Actual)
Dates: Start 2000-11; Primary Completion 2002-08 (Actual); Study Completion 2002-08 (Actual)

PRIMARY OUTCOMES:
Time to meet discharge criteria (functional airway improvement)during the first 3 hours of Period I. | 24 hours

SECONDARY OUTCOMES:
FEV1 (Period I): Serial spirometry, maximum FEV1, time to maximum FEV1, baseline FEV1 severity on subject response; % responders, no. nebulizations to meet discharge criteria, rate of hospitalization, time to admit decision, rate for increased care | Day 0 (5-10 min after every dose)
FEV1 (Period II): Spirometry, average FEV1; distribution of subject responses; rate of relapse; blinded study medication; length of stay in ED or Clinic during Period I; length of hospitalization, cost of care | Days 3, 10
Investigator and subject global evaluations, subject preference | Days 3, 10
Subject reported beta-mediated side effects | Days 3, 10

CONTACTS AND LOCATIONS:
Locations (28):
- United States (28):
  - Hoover, Alabama
  - Montgomery, Alabama
  - Encinitas, California
  - Fresno, California
  - Oakland, California
  - Torrance, California
  - Colorado Springs, Colorado
  - Gainesville, Florida
  - Jacksonville, Florida
  - Tampa, Florida
  - Chicago, Illinois
  - Metairie, Louisiana
  - Ann Arbor, Michigan
  - Detroit, Michigan
  - Kansas City, Missouri
  - St Louis, Missouri
  - Red Bank, New Jersey
  - Brooklyn, New York
  - New Hyde Park, New York
  - Syracuse, New York
  - Rocky Mount, North Carolina
  - Akron, Ohio
  - Cleveland, Ohio
  - Lake Oswego, Oregon
  - Medford, Oregon
  - Philadelphia, Pennsylvania
  - Houston, Texas
  - Salt Lake City, Utah